CLINICAL TRIAL: NCT04189692
Title: Evolution of Fatigue in Patients With Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Diana Horta-Sangenis, gastroenterologist physician, Corporacion Parc Tauli
Other Study IDs: HMT3
Record Dates: First submitted 2019-11-14; First posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Fatigue; Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: Fatigue;; Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Fatigue; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Inflammatory Bowel Disease and fatigue: Patients with Inflammatory Bowel Disease and fatigue that participated in the two studies (1,2).

SUMMARY:
The aim of this study is to evaluate the evolution and possible factors associated with the persistence of fatigue in patients with quiescent IBD and fatigue included in two previous studies.

DETAILED DESCRIPTION:
Fatigue is a common symptom in inflammatory bowel disease and persists despite clinical remission. Fatigue in patients with chronic diseases can be objectified by the FACIT-F scale.

Recent publications have tried to assess the prevalence and factors related to fatigue in patients with IBD.

In 2017 one study evaluated the prevalence and predictive factors of fatigue in out-patients with inflammatory bowel disease. Fatigue was associated with depression, low quality of life and female sex. No association was found with micronutrients or levels of interleukins.

As there are no effective treatments for fatigue in IBD, another study, recently published a study evaluating the role of electroacupuncture in 54 patients with quiescent IBD and fatigue, observing that both electroacupuncture and sham acupuncture improved fatigue compared to the control group.

The aim of this study is to evaluate the evolution and possible factors associated with the persistence of fatigue in patients with quiescent IBD and fatigue included in the two previous studies.

Patients with inflammatory bowel disease and fatigue (FACIT-F score < 40) included in these two previous studies who agree to participate will fill in questionnaires to assess fatigue, anxiety, depression and quality of life in inflammatory bowel disease. Moreover, the relationship of other biological factors with IBD-related fatigue will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease and fatigue (defined as a FACIT-F score <40 points) previously documented in our two previous studies.
* Written informed consent after receiving clear and objective information about the purpose and characteristics of the study.
* Ability to understand the questionnaires.

Exclusion Criteria:

* Associated tumor disease.
* Pregnancy or breastfeeding.
* Anemia (hemoglobin <12g/dl in women and 14g/dl in men)
* Any concomitant illness that may justify the presence of fatigue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with IBD and fatigue included in the two previous studies (1,2) (n = 202) who agree to participate.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2020-01-07 (Estimated); Primary Completion 2020-12-07 (Estimated); Study Completion 2020-12-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the evolution of fatigue in patients with Inflammatory Bowel Disease at 3 years | three years
  Assessed by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F scale). This questionnaire, previously validated in Spanish and for IBD patients, comprises 40 items divided into five subscales: Physical wellbeing (PWB), Social/family wellbeing (SWB), Emotional wellbeing (EWB), Functional Wellbeing (FWB), and Fatigue subscale. The first four subscales (27 items) evaluate general features of chronic illness, and the 13 items of the Fatigue subscale specifically focus on fatigue. Each item has five possible answers, from 0 (very fatigued) to 4 (not at all fatigued). The score of each subscale is the sum of the coded values of its items.

SECONDARY OUTCOMES:
Assess the biological factors associated with the persistence of fatigue | three years
  Assessed by a blood test including micronutrients (vitamin B12, ferritin and vitamin D).
Assess the psychological factors associated with the persistence of fatigue | three years
  Assessed by the Beck Depression Inventory (BDI) questionnaire. The Spanish validated 21-item version of the BDI will be used to analyze depression. This self-administered questionnaire evaluates the clinical features of melancholy and intrusive thoughts present in depression. Each item has a different number of options (from 4 to 8), which then have to be converted into four possible values (0, 1, 2, or 3). Higher BDI scores indicate a higher grade of depression.
Assess the psychological factors associated with the persistence of fatigue | three years
  Assessed by Quality of life in inflammatory bowel disease questionnaire (IBDQ-9). he IBDQ-9 consists of nine items assessing different aspects of life in IBD patients. Each item has seven different possible answers, scoring from 1 (poorest) to 7 (best). The straight summation of all nine items provides a direct score, which is then transformed into a final score. Higher scores correspond to a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Horta, Principal Investigator — Parc Tauli Hospital. Sabadell , Barcelona, Spain, 08208

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villoria A, Garcia V, Dosal A, Moreno L, Montserrat A, Figuerola A, Horta D, Calvet X, Ramirez-Lazaro MJ. Fatigue in out-patients with inflammatory bowel disease: Prevalence and predictive factors. PLoS One. 2017 Jul 27;12(7):e0181435. doi: 10.1371/journal.pone.0181435. eCollection 2017. PMID 28749985
- [Background] Horta D, Lira A, Sanchez-Lloansi M, Villoria A, Teggiachi M, Garcia-Rojo D, Garcia-Molina S, Figuerola A, Esteve M, Calvet X. A Prospective Pilot Randomized Study: Electroacupuncture vs. Sham Procedure for the Treatment of Fatigue in Patients With Quiescent Inflammatory Bowel Disease. Inflamm Bowel Dis. 2020 Feb 11;26(3):484-492. doi: 10.1093/ibd/izz091. PMID 31091322